CLINICAL TRIAL: NCT02611856
Title: STT Study : Pediatric Follow-up of Children's From Monochorial-diamniotic Pregnancies Complicated With a Twin-to-twin Syndrome
Brief Title: Monochorial-diamniotic Pregnancies Complicated With a Twin-to-twin Syndrome
Acronym: STT
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Société Française d'Hypentension Artérielle (Other)
Responsible Party: Sponsor
Other Study IDs: CRC05069
Record Dates: First submitted 2015-07-02; First posted 2015-11-23 (Estimated); Last update posted 2021-07-07 (Actual); Status verified 2021-06

CONDITIONS: Twin to Twin Transfusion Syndrome
Keywords: twin to twin,; transfusion syndrome
MeSH Terms: conditions — Fetofetal Transfusion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — sera, urine
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- monochorial-biamniotic pregnancies

SUMMARY:
The twin pregnancies monochorionic are specifically explained to two main types of complications: the anomalies of the embryo affecting a symmetry and in particular the median line on one hand and malformative sequences of vascular origin on the other hand. This last category of anomalies (twin-to-twin syndrome, TTTS) develops because of the presence of a division of the foeto-placentary circulation between both twins through the pooling of certain placentary cotyledons. The latter are then vascularized by an arterial and venous foot belonging to both foetuses (anastomoses arteria-venous or veinous-arterial). It results from it an imbalance moderate but very early hemodynamic which is going to return a hypovolume twin (the donor) and its plethoric co-twin (the recipient).

These anomalies in utero could not only have consequences during the fetal life, on the born weight and the later development of newborns, but also on the organization and the functioning of a whole series of physiological systems. So these anomalies of the pregnancy could have also consequences which exceed by very far from the perinatal period, by favoring the development of the atheroma, the high blood pressure, the resistance in the insulin, and many other metabolic and endocrine functions were known for their importance in human pathology.

For these reasons the investigators suggest estimating the tensional, cardiac and metabolic status of children ex-transfusers and of children ex-transfused in 2 different age classes: between 4 and 8 years then when these children will have between 12 and 16 years.

There are also some evaluation clinical and biological of the puberty (only at the age of 12-16)

To understand a possible effect of the prenatal status of these children on the endocrinology of the puberty, the measures and the following dosages will be realized:

* Test in the GnRH (T0, T30, T60, T90): dosages of LH and FSH (relationship of peaks to determine the puberty evolution),
* Dosages of the sexual steroids, the oestradiol for the girl and the testosterone for the boy,
* Clinical examination looking for the signs of puberty

This if study leans on the big originality of the physiopathological model of TTTS in which the children present the peculiarity to have an identical genetic and postnatal status and a different prenatal environment.

The follow-up of these children should allow:

* To understand better the postnatal impact anomalies on these children in the course of pregnancy
* To anticipate and thus to improve their care in case of appearance of biological or clinical signs

ELIGIBILITY:
Inclusion Criteria:

* Child (ren) from (s) of a twin pregnancy with fetal transfusion syndrome fetal
* Child (ren) age (s) 4 years 0 months to 6 years 12 months
* Child (ren) fasting
* Consent signed by the parents or legal representative

Exclusion Criteria:

* Child (ren) not derived (s) of a twin pregnancy with fetal transfusion syndrome fetal
* Child (ren) age (s) under 4 years 0 months or more than 6 years 12 months
* Child (ren) nonfasting

Ages: 4 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children aged 4 years to 8 years
Sampling Method: Non-Probability Sample
Enrollment: 179 (Actual)
Dates: Start 2007-04-03 (Actual); Primary Completion 2022-06-30 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Composite measure of the cardiac function | one day
  * measure of the arterial blood pressure
  * cardiac echography
Composite measure of the renal function | one day
  * microalbuminuria
  * level of plasmatic renin, plasmatic cortisol, prorenin, aldosterone
  * renal echography

SECONDARY OUTCOMES:
Composite measure of the glycoregulation | one day
  * provoked oral hyperglycemia
  * level of glycemia
  * level of insulinemia
  * level of glycosuria

CONTACTS AND LOCATIONS:
Overall Officials: Laurence Bussières, Ph.D, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hôpital Robert Debré, Paris, France